CLINICAL TRIAL: NCT02970370
Title: Demographics, Clinical and Paraclinical Characteristics of Multiple Sclerosis in Egypt
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hatem Samir Shehata, Professor of Neurology, Cairo University
Other Study IDs: Cairo-5-UMP
Record Dates: First submitted 2016-11-18; First posted 2016-11-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 15 Years

INTERVENTIONS:
Other: no intervention

SUMMARY:
The primary study aim is to depict the demographics, clinical and para clinical features of patients attending five tertiary referral multiple sclerosis (MS) centers in Egypt.

This requires effective and unified pooled registries to extract data from with a standardized, sufficient and high quality clinical, magnetic resonance imaging (MRI) data, neurophysiological data and body fluids.

Investigators want to shed light on the challenges that face both physicians and patients in the area of "diagnosis and treatment"

ELIGIBILITY:
Inclusion Criteria:

* Patients with MS/NMOSD or their mimics who sought advice in one of our centers even once

Exclusion Criteria:

* Patients with missing data in their records that couldn't be completed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Radiologically isolated syndrome, Clinically isolated Syndrome , Multiple Sclerosis, Neuromyelitis optica spectrum disorders (NMOSD), MS mimics
Sampling Method: Non-Probability Sample
Enrollment: 2752 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
portrayed phenotypes and para-clinical data of Egyptian Multiple Sclerosis Patients | 6 months